CLINICAL TRIAL: NCT01435954
Title: Clinical Progression and Costs in Benign Prostatic Hyperplasia Patients Treated With Early Versus Delayed Combination Therapy
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 113908
Record Dates: First submitted 2011-09-15; First posted 2011-09-19 (Estimated); Last update posted 2017-05-16 (Actual); Status verified 2017-05

CONDITIONS: Benign Prostatic Hyperplasia
Keywords: benign prostatic hyperplasia; surgery; 5-alpha-reductase inhibitor; enlarged prostate; acute urinary retention
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with Benign Prostatic Hyperplasia (BPH): Insured male patients age 50 or older with BPH but no evidence of acute urinary retention (AUR) or prostate surgery at the index date
  Interventions: Drug: Early combination therapy; Drug: Delayed combination therapy

INTERVENTIONS:
Drug: Early combination therapy — If index drug was an alpha-blocker (AB) (alfuzosin, doxazosin, tamsulosin, or terazosin), a pharmacy claims for a 5-alpha reductase inhibitor (5ARI) (dutasteride, finasteride) on or within 30 days after the index date or if index drug was 5ARI, fill for an AB on or within 30 days after the index date
  Other Names: Flomax® is a registered trademark of Astellas Pharma; Rapaflo® is a registered trademark of Watson Pharmaceuticals; Inc; Proscar® is a registered trademark of Merck; Uroxatral® is a registered trademark of Sanofi-Aventis; Cardura® is a registered trademark of Pfizer Inc; Avodart® is a registered trademark of GlaxoSmithKline; Hytrin® is a registered trademark of Abbott Laboratories
Drug: Delayed combination therapy — If index drug was an AB (alfuzosin, doxazosin, tamsulosin, or terazosin), a pharmacy claim for a 5ARI (dutasteride, finasteride) more than 30 days but less than or equal to 180 days of the index date
  Other Names: Cardura® is a registered trademark of Pfizer Inc; Proscar® is a registered trademark of Merck; Hytrin® is a registered trademark of Abbott Laboratories; Uroxatral® is a registered trademark of Sanofi-Aventis; Avodart® is a registered trademark of GlaxoSmithKline; Rapaflo® is a registered trademark of Watson Pharmaceuticals; Inc; Flomax® is a registered trademark of Astellas Pharma

SUMMARY:
In patients with benign prostatic hyperplasia (BPH), combination therapy with an alpha-blocker (AB) and a 5 alpha-reductase inhibitor (5ARI) has been shown to reduce the progression of acute urinary retention (AUR) and the incidence of prostate surgery, and also provides symptom relief.

The objective of this study is to compare the likelihood of clinical progression (defined as AUR and/or prostate-related surgery) and costs in BPH patients who were treated with delayed combination therapy to BPH patients who were treated with early combination therapy using data from a United States (US) healthcare claims database. The hypothesis of this study is that patients who are prescribed combination therapy early in their BPH treatment will experience better clinical outcomes and lower healthcare costs compared with patients treated with delayed combination therapy. The null hypothesis is that no difference will be observed in outcomes or direct medical costs for patients treated with early combination therapy and patients treated with delayed combination therapy.

The US healthcare claims database includes data from patients with Medicare Advantage as well as private health plan coverage including the Impact health plan. About 14 million people were covered by this set of health plans in 2007 and were geographically diverse across the US. Data from 2000 through 2009 were utilized.

The study is a retrospective cohort analysis.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Age 50 or older at the index date (the date of the first filled prescription for an AB or 5ARI during the enrollment period)
* At least one claim with an ICD-9 diagnosis code for BPH (222.2 or 600.xx) in any position and at least one pharmacy claim for an AB (alfuzosin, doxazosin, tamsulosin, or terazosin) or at least one fill for a 5ARI (dutasteride or finasteride) (with or without a diagnosis for BPH)
* Continuous enrollment with medical and pharmacy benefits for 6 months prior to the index date (i.e., baseline period) and 12 months after the index date (follow-up period)

Exclusion Criteria:

* At least one pharmacy claim for an AB (alfuzosin, doxazosin, tamsulosin, or terazosin) any time during the pre-index period prior to the index date
* At least one fill for a 5ARI (dutasteride or finasteride) any time during the pre-index period prior to the index date
* A diagnosis code for prostate cancer (ICD-9 = 185, 198.82, 233.4, 236.5, 239.5, V10.46) or bladder cancer (ICD-9 =188, 198.1, 223.3, 233.7, 239.4, V10.51) in any position during the pre-index or follow-up period
* A pharmacy claim for finasteride 1 mg tablets (i.e., treatment of male-pattern baldness) during the pre-index or follow-up period
* Prostate surgery anytime during the pre-index period or 5 months after the index date

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Insured male patients, aged 50 and older, with a diagnosis of benign prostatic hyperplasia (BPH) as identified by International Classification of Diseases, 9th Revision, Clinical Modification (ICD-9) codes for BPH (ICD-9 = 222.2x or 600.xx)
Sampling Method: Non-Probability Sample
Enrollment: 13551 (Actual)
Dates: Start 2010-08; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Number of participants with a code that indicates clinical progression | Data collected over a 9-year time period from 2000 to 2009.
  The number of participants who experience clinical progresion (BPH-surgery or AUR) based on treatment or diagnosis codes and compared between participant records of BPH patients treated with early combination therapy compared with delayed combination therapy

SECONDARY OUTCOMES:
Mean BPH-related medical costs | Data collected over a 9-year time period from 2000 to 2009
  The mean cost of medical treatment related to BPH in US dollars for records of patients who were treated with early combination therapy and those treated with delayed combination therapy

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline